CLINICAL TRIAL: NCT03739450
Title: Problem Solving Training for Care Partners of Adults With Traumatic Brain Injury
Acronym: CP-PST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Baylor Health Care System (Other); Kessler Institute for Rehabilitation (Industry); Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, Shannon Juengst, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 042018-052; 90DPTB0013-01-00 (Other Grant/Funding Number: Other)
Record Dates: First submitted 2018-11-01; First posted 2018-11-13 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Care Partners of Patients With Traumatic Brain Injury (TBI)
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants are randomized and allocated after baseline assessment to PST + Education or Education only via stratified, blocked randomization. Randomization is stratified by participating center and then based on whether a single care partner or multiple care partners are participating for the same patient by participating TBIMS Center. The investigators used a block size of four to ensure equal numbers across groups and to account for potentially small numbers of participants at any given TBIMS Center. Randomization is computer-generated and maintained by the TBI Model Systems National and Statistical Data Center. Allocation assignments for each center are distributed to the site PI and maintained in a password-protected electronic file. Outcome assessors are blinded to intervention allocation.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be ensured by allocating to group assignment after baseline assessment is complete, having different staff performing assessments vs delivering the intervention, scheduling meetings with assessors and interventionists separately, and instructing participants to not discuss the intervention with the person calling to complete follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Solving Training + Education (Experimental): Participants in this arm will receive the TBI-specific education intervention and the Problem Solving Training (PST) intervention.
  Interventions: Behavioral: Problem Solving Training (PST); Behavioral: Education
- Education (Active Comparator): Participants in this arm will only receive the TBI-specific education intervention.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Problem Solving Training (PST) — The PST intervention consists of six sessions that will follow a structured format based on the PST manual. In these sessions, the interventionist will first provide the TBI-specific education, introduce the participant to the PST steps, then help the care partner generate and select a problem to address first. Interventionist will facilitate the care partner's use of the ABCDEF steps of PST to develop a specific action plan to solve the problem. As problems are attempted or solved, the care partner will learn how to perform the steps on his/her own, thus acquiring self-management problem solving skills that will be applicable to future problems. The final session will include a review and generalization of the PST steps and progress made.
  Arms: Problem Solving Training + Education
Behavioral: Education — Participants will receive TBI-specific education alone through a workbook. It consists of educational modules for self-study, common sequelae of TBI, issues encountered by care partners, work and school concerns for those with TBI, and on navigating the rehab system and accessing resources. The modules consist of a brief introduction, key definitions, examples, resources, and a summary. Some chapters also include self-directed activities, such as worksheets or checklists. The investigators will provide a brief orientation to the workbook and include open-ended questions about the participants' need for clarification or questions of the education material. The last session will consist of an open discussion about expected problems that may arise post-discharge.

SUMMARY:
Importance: The chronic consequences of TBI are established, but ongoing support for adults with TBI living in the community is limited. This puts undue burden on care partners, particularly during the transition from hospital to home. It often leads to adverse consequences among care partners, such as emotional distress and increased substance abuse. Currently, there are no evidence-based interventions for care partners of adults with TBI to prepare them for this role. Problem Solving Training (PST) is an evidence-based, self-management approach with demonstrated efficacy for care partners of individuals with disabilities, but it has not been delivered or evaluated during inpatient rehabilitation.

Aims: Aim 1): To assess the feasibility of providing PST to care partners of adults with TBI during the inpatient rehabilitation stay; Aim 2) To assess the efficacy of PST + education vs education alone for improving caregiver burden, depressive symptoms, and coping skills Method: The investigators will conduct a randomized control trial of PST + Education vs Education alone during the inpatient rehabilitation stay of individuals with TBI. The investigators will enroll 172 care partners and conduct baseline assessment, with follow-up assessment at 1 month and 6 months post-discharge. For Aim 1, the investigators will measure number of sessions of PST completed and care partner satisfaction. For Aim 2, the investigators will compare differences in PST+Educaion vs. Education alone in measures of caregiver burden, depressive symptoms, and coping skills at 1-month and 6-months post-discharge.

Conclusion: The investigators anticipate that care partners will be able to complete a minimum of 3 sessions during the inpatient rehabilitation stay and that PST + Education will be more effective than Education alone for reducing caregiver burden and depressive symptoms and improving positive coping among care partners. PST is an evidence-based, self-management approach with a strong theoretical foundation that has demonstrated efficacy for care partners of individuals with disabilities. Early work indicates that it is also effective for care partners of adults with TBI. However, there are no studies evaluating whether delivery of PST to care partners is feasible during inpatient rehabilitation. The proposed project builds upon this foundation of evidence to address this critical gap in the literature. It will provide evidence for effective ways to support and improve outcomes for care partners during the transition from hospital to home.

DETAILED DESCRIPTION:
North TX TBIMS Module Project: Problem Solving Training (PST) for Care Partners of Adults with Traumatic Brain Injuries (TBI) during Inpatient Rehabilitation

Care partners of adults with TBI report substantial burden and emotional distress and a need for more resources and skills training to manage the transition from hospital to home.

The investigators will assess the feasibility and efficacy of Problem Solving Training for care partners during inpatient rehabilitation to reduce burden and depressive symptoms and improve coping across the critical transition from inpatient rehabilitation to the community.

Statement of Problem: The chronic consequences of TBI are recognized, but ongoing support for adults with TBI living in the community is limited. This puts undue burden on care partners, particularly during the transition from hospital to home. It often leads to adverse consequences among care partners, such as emotional distress and increased substance abuse.1,2 Care partners of individuals with TBI often experience high levels of burden, which may result in depression, anxiety, increased somatic symptoms, and reduced quality of life.1,3,4 Care partner burden is largely predicted by the extent to which care partners' perceived needs are met.1,5,6 As the consequences of TBI continue to change over time, so too do the perceived needs of care partners.7-11 One study suggests that only 55% of care partner needs are perceived as being met.12 A systematic review of qualitative studies for care partners of adults with stroke revealed seven themes with regard to experiences, needs, and preferences of care partners during inpatient rehabilitation.13 Care partners expressed a desire to be included, informed, and recognized as a stakeholder in recovery, the need to navigate an alien culture and environment, and the need to manage the transition home.13 The authors concluded that "the investigators need to make deliberate efforts to provide a more inclusive environment that better supports and prepares carers for their new role".13 Despite this established need during inpatient rehabilitation, there are currently no evidence-based interventions for care partners of adults with TBI to prepare them for their new role prior to discharge of care recipients from inpatient rehabilitation. Hence, there is a critical need to provide care partners of individuals with TBI with the necessary skills to navigate this difficult transition from hospital to home.14 Self-management training for care partners of adults with other chronic conditions demonstrates strong potential for application to care partners of adults with TBI.

Proposed Solution: Problem-Solving Training (PST) is an evidence-based, self-management approach that teaches a simple, systematic method for evaluating problems, generating and selecting solutions, creating and implementing realistic goals and action plans, and evaluating whether those plans effectively addressed the specific goal.15,16 A growing body of evidence indicates that PST post-discharge is associated with reduced distress among care partners of adults with TBI.17-19 Problems previously seen as overwhelming are regarded as solvable and manageable when approached in a stepwise fashion using PST, thereby reducing perceived burden and emotional distress. PST empowers care partners to be active participants in directing health and rehabilitation services.

Specific Aims:

Specific Aim 1: To assess the feasibility (compliance, satisfaction) of delivering Problem Solving Training (PST) to care partners of individuals with TBI during inpatient rehabilitation.

Specific Aim 2: To assess the efficacy of PST plus TBI-specific education compared to TBI-specific education alone for improving the outcomes of care partners of individuals with TBI.

Method: The investigators will conduct a randomized control trial of PST + Education vs Education alone during the inpatient rehabilitation stay of individuals with TBI. The investigators will enroll 172 care partners across sites and conduct baseline assessment, with follow-up assessment at 1 month and 6 months post-discharge.

Sample size: The investigators plan to enroll 172 care partners to achieve an effect size (group differences in burden at 1 month) of Cohen's d=.40; α=0.05, power=80%, and attrition=10%. With recruitment projected to occur for 27 months, this would require recruiting 6-7 participants per month across participating sites.

Description of Intervention: Care partners in the intervention group will receive PST training plus TBI-specific education (6 sessions). Participants in the Control group will receive TBI-specific education alone (6 points of contact).19 Sessions will last ~30-60 minutes each. All sessions will occur in-person whenever possible, or over the telephone when meeting is not feasible. PST has been successfully delivered via both modalities, with similar effects. Our group has particular experience delivering PST via telephone.19-22 Control group points of contact for education will last ~15 minutes each, with the first and last session conducted in person and other contacts by phone. Trained members of the research team with master's level education or equivalent experience will provide both interventions using a specific curriculum that has been validated in our previous research studies20. These activities will take place before discharge from inpatient rehabilitation. A structured database will be used to record the session delivery to ensure fidelity, including completion, reasons for non-compliance, method of delivery, session length, and a brief summary of the PST steps covered during session.

Assessments: For Aim 1, the investigators will measure number of PST sessions completed, if a minimum of 3 sessions were completed (Y/N), and care partner satisfaction. For Aim 2, the investigators will compare differences in PST+Education vs. Education alone in measures of caregiver burden, depressive symptoms, and coping skills, including alcohol use, at 1-month and 6-months post-discharge. The investigators will explore sustainability of the PST intervention at 6-months, testing group by time interactions for caregiver burden, depressive symptoms, and coping. Outcomes measures will include the Alcohol Use Disorders Identification Test (AUDIT),23 Brief Coping Orientation to Problems Experienced (Brief COPE),24 Patient Health Questionnaire 9 (PHQ9),25 Zarit Burden Interview (ZBI),26 and the Client Satisfaction Questionnaire (CSQ8).27 Analysis Plan: The primary outcome to assess feasibility is the completion of a minimum of 3 sessions of PST. The investigators will also report the number of sessions completed prior to discharge, and method of completion (in person or via telephone), to inform future intervention design. The investigators will descriptively present reasons for non-compliance, captured through our intervention database. The investigators will divide the participants into two groups, based upon completion of <3 sessions or >3 sessions. The investigators will then compare the two groups and explore demographic or other baseline differences (e.g. in outcomes of interest, in inpatient length of stay, etc.) to identify factors associated with compliance. The investigators will compare the level of client satisfaction (CSQ-8) with the intervention in both groups. For all group comparisons, the investigators will use t-tests, Mann-Whitney U test, or Chi Squared tests, as appropriate.

The investigators will calculate measures of central tendency or numbers and percentages for all demographic baseline variables and descriptively compare PST Intervention to Education groups, to reduce the overall number of comparisons and the likelihood of a type I error. If there are group differences, the investigators will conduct formal statistical testing (t-tests, Mann Whitney U tests, or Chi Square tests, as appropriate) to determine potential confounding variables resulting from initial group differences and adjust for these variables accordingly. The investigators will use intent-to-treat analyses to measure the differences in each outcome measure between PST Intervention vs. Education groups at 1-month follow-up using t-tests or Mann Whitney U tests, as appropriate. If covariate adjustment is determined to be necessary based on baseline differences between the two groups, the investigators will conduct Analysis of Covariance (ANCOVA) for each outcome, adjusting for relevant factors. To address our second hypothesis, the investigators will assess group by time interactions, including baseline, 1-month, and 6-month time points, using repeated-measures ANOVA/ANCOVA. For the coping skills outcome, the investigators will use baseline data from all participants and conduct exploratory factor analysis to identify second-order factors in our sample as a means of data reduction and analyze total scores within the second-order factors.

Implementation of research design is feasible given the time and resources: The investigators have previously conducted a RCT delivering PST to 77 care partners of adults with TBI via telephone beginning one week post-discharge.19 Care partners completed up to 10 sessions, with 8 sessions as a target. Of the 77 participants, 41 (53.2%) completed 7-10 sessions, 30 (39.0%) completed 1-6 sessions, and 6 (7.8%) did not complete any sessions after randomization. Dr. Juengst has experience as a treating therapist, trainer, and supervisor for self-management interventions, including assessing treatment fidelity and navigating intervention delivery during inpatient rehabilitation. She will train participating centers in the conduct of this project via webinar and using a written manual. Interventionists will demonstrate competency in the intervention before use. Assessments are self-reported, can be completed by a research assistant (blinded to intervention allocation), and take 20-30 minutes to complete. Our timeline is feasible based on our past experience recruiting participants, delivering self-management interventions, and participating in TBIMS modules Addition to State-of-the-Art: The investigators anticipate that care partners will be able to complete a minimum of 3 sessions during the inpatient rehabilitation stay, with the goal of completing 6 sessions. The investigators also anticipate that PST + Education will be more effective than Education alone for reducing caregiver burden and depressive symptoms and improving positive coping among care partners. This study will provide evidence for effective strategies to support and improve outcomes for care partners during the transition from hospital to home. This will benefit the TBIMS as a whole by providing an evidence-based and feasible intervention for care partners, upon whom the TBIMS relies heavily for participant enrollment and data collection, in addition to the ongoing support that care partners provide to the primary beneficiaries of TBIMS services, individuals with TBI. PST is an evidence-based, self-management approach with a strong theoretical foundation that has demonstrated efficacy for care partners of individuals with disabilities. Early work indicates that it is also effective for care partners of adults with TBI. However, there are no studies evaluating whether delivery of PST to care partners is feasible and effective during inpatient rehabilitation. The proposed project builds upon this foundation of evidence to address this critical gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Identified as care partner of an individual with TBI admitted to inpatient rehabilitation. A care partner is defined as an individual (spouse, partner, family member, friends, or neighbor) involved in assisting the patient with activities of daily living and/or medical tasks or responsible in any way for the patient's well-being after discharge from inpatient rehabilitation.
2. >1-year relationship
3. Ability to communicate in English.
4. >18 years old
5. Capacity to self-consent

Exclusion Criteria:

Dispute over care partner's role in the care of patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Juengst, PhD, Principal Investigator — UT Southwestern
Locations (4):
- United States (4):
  - Kessler Foundation, East Hanover, New Jersey
  - JFK Johnson Rehabilitation Institute, Edison, New Jersey
  - Baylor Scott & White Institute for Rehabilitation, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The IPD that will be shared includes the study protocol, the statistical analysis plan and the clinical study report.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The research module data will remain under the control of the lead project team for one year after completion of data collection of the project. This will allow ample time for analyses and preparation of planned manuscripts. After the one-year period, any of the centers may request the data for additional analysis and dissemination. See SOP 6b for more details on internal procedures.
Access Criteria: Both internal and external entities may request IPD through two separate procedures.
  Internal Use:
  Participating site in the TBI Model Systems may reference SOP 602b for further procedures.
  External Use:
  All staff, students, and other related personnel not involved in the NIDILRR-funded TBI Model Systems Centers or Follow-up Centers who wish to use data from the TBI Model Systems National Database or Modules may request access to the data set by completing a Data Request and Use Agreement Form available for download at www.tbindsc.org The Data Request and Use Agreement Form, once complete, can be emailed or faxed to the Project Director of the TBI Model Systems National Data and Statistical Center (see www.tbindsc.org and go to contacts).
  Reference: SOP 602d

REFERENCES:
- [Background] Manskow US, Sigurdardottir S, Roe C, Andelic N, Skandsen T, Damsgard E, Elmstahl S, Anke A. Factors Affecting Caregiver Burden 1 Year After Severe Traumatic Brain Injury: A Prospective Nationwide Multicenter Study. J Head Trauma Rehabil. 2015 Nov-Dec;30(6):411-23. doi: 10.1097/HTR.0000000000000085. PMID 25119652
- [Background] Bayen E, Jourdan C, Ghout I, Darnoux E, Azerad S, Vallat-Azouvi C, Weiss JJ, Aegerter P, Pradat-Diehl P, Joel ME, Azouvi P. Objective and Subjective Burden of Informal Caregivers 4 Years After a Severe Traumatic Brain Injury: Results From the PariS-TBI Study. J Head Trauma Rehabil. 2016 Sep-Oct;31(5):E59-67. doi: 10.1097/HTR.0000000000000079. PMID 24992640
- [Background] Kreutzer JS, Gervasio AH, Camplair PS. Primary caregivers' psychological status and family functioning after traumatic brain injury. Brain Inj. 1994 Apr;8(3):197-210. doi: 10.3109/02699059409150973. PMID 8004079
- [Background] Kolakowsky-Hayner SA, Miner KD, Kreutzer JS. Long-term life quality and family needs after traumatic brain injury. J Head Trauma Rehabil. 2001 Aug;16(4):374-85. doi: 10.1097/00001199-200108000-00007. PMID 11461659
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Davis LC, Sander AM, Struchen MA, Sherer M, Nakase-Richardson R, Malec JF. Medical and psychosocial predictors of caregiver distress and perceived burden following traumatic brain injury. J Head Trauma Rehabil. 2009 May-Jun;24(3):145-54. doi: 10.1097/HTR.0b013e3181a0b291. PMID 19461362
- [Background] Kreutzer JS, Gervasio AH, Camplair PS. Patient correlates of caregivers' distress and family functioning after traumatic brain injury. Brain Inj. 1994 Apr;8(3):211-30. doi: 10.3109/02699059409150974. PMID 8004080
- [Background] Ponsford J, Olver J, Ponsford M, Nelms R. Long-term adjustment of families following traumatic brain injury where comprehensive rehabilitation has been provided. Brain Inj. 2003 Jun;17(6):453-68. doi: 10.1080/0269905031000070143. PMID 12745702
- [Background] Nabors N, Seacat J, Rosenthal M. Predictors of caregiver burden following traumatic brain injury. Brain Inj. 2002 Dec;16(12):1039-50. doi: 10.1080/02699050210155285. PMID 12487718
- [Background] Rotondi AJ, Sinkule J, Balzer K, Harris J, Moldovan R. A qualitative needs assessment of persons who have experienced traumatic brain injury and their primary family caregivers. J Head Trauma Rehabil. 2007 Jan-Feb;22(1):14-25. doi: 10.1097/00001199-200701000-00002. PMID 17235227
- [Background] Murphy MP, Carmine H. Long-term health implications of individuals with TBI: a rehabilitation perspective. NeuroRehabilitation. 2012;31(1):85-94. doi: 10.3233/NRE-2012-0777. PMID 22523016
- [Background] Lefebvre H, Levert MJ. The close relatives of people who have had a traumatic brain injury and their special needs. Brain Inj. 2012;26(9):1084-97. doi: 10.3109/02699052.2012.666364. Epub 2012 May 24. PMID 22624724
- [Background] Luker J, Murray C, Lynch E, Bernhardsson S, Shannon M, Bernhardt J. Carers' Experiences, Needs, and Preferences During Inpatient Stroke Rehabilitation: A Systematic Review of Qualitative Studies. Arch Phys Med Rehabil. 2017 Sep;98(9):1852-1862.e13. doi: 10.1016/j.apmr.2017.02.024. Epub 2017 Mar 28. PMID 28363703
- [Background] Gan C, Gargaro J, Brandys C, Gerber G, Boschen K. Family caregivers' support needs after brain injury: a synthesis of perspectives from caregivers, programs, and researchers. NeuroRehabilitation. 2010;27(1):5-18. doi: 10.3233/NRE-2010-0577. PMID 20634597
- [Background] Malouff JM, Thorsteinsson EB, Schutte NS. The efficacy of problem solving therapy in reducing mental and physical health problems: a meta-analysis. Clin Psychol Rev. 2007 Jan;27(1):46-57. doi: 10.1016/j.cpr.2005.12.005. Epub 2006 Feb 9. PMID 16480801
- [Background] Grant JS, Elliott TR, Weaver M, Bartolucci AA, Giger JN. Telephone intervention with family caregivers of stroke survivors after rehabilitation. Stroke. 2002 Aug;33(8):2060-5. doi: 10.1161/01.str.0000020711.38824.e3. PMID 12154263
- [Background] Rivera PA, Elliott TR, Berry JW, Grant JS. Problem-solving training for family caregivers of persons with traumatic brain injuries: a randomized controlled trial. Arch Phys Med Rehabil. 2008 May;89(5):931-41. doi: 10.1016/j.apmr.2007.12.032. PMID 18452743
- [Background] Powell JM, Fraser R, Brockway JA, Temkin N, Bell KR. A Telehealth Approach to Caregiver Self-Management Following Traumatic Brain Injury: A Randomized Controlled Trial. J Head Trauma Rehabil. 2016 May-Jun;31(3):180-90. doi: 10.1097/HTR.0000000000000167. PMID 26394294
- [Background] Bell KR, Brockway JA, Fann JR, Cole WR, St De Lore J, Bush N, Lang AJ, Hart T, Warren M, Dikmen S, Temkin N, Jain S, Raman R, Stein MB. Concussion treatment after combat trauma: development of a telephone based, problem solving intervention for service members. Contemp Clin Trials. 2015 Jan;40:54-62. doi: 10.1016/j.cct.2014.11.001. Epub 2014 Nov 8. PMID 25460344
- [Background] Bell KR, Fann JR, Brockway JA, Cole WR, Bush NE, Dikmen S, Hart T, Lang AJ, Grant G, Gahm G, Reger MA, St De Lore J, Machamer J, Ernstrom K, Raman R, Jain S, Stein MB, Temkin N. Telephone Problem Solving for Service Members with Mild Traumatic Brain Injury: A Randomized, Clinical Trial. J Neurotrauma. 2017 Jan 15;34(2):313-321. doi: 10.1089/neu.2016.4444. Epub 2016 Oct 13. PMID 27579992
- [Background] Bell KR, Brockway JA, Hart T, Whyte J, Sherer M, Fraser RT, Temkin NR, Dikmen SS. Scheduled telephone intervention for traumatic brain injury: a multicenter randomized controlled trial. Arch Phys Med Rehabil. 2011 Oct;92(10):1552-60. doi: 10.1016/j.apmr.2011.05.018. PMID 21963122
- [Background] Bryce S, Spitz G, Ponsford J. Screening for Substance Use Disorders Following Traumatic Brain Injury: Examining the Validity of the AUDIT and the DAST. J Head Trauma Rehabil. 2015 Sep-Oct;30(5):E40-8. doi: 10.1097/HTR.0000000000000091. PMID 25310295
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Fann JR, Bombardier CH, Dikmen S, Esselman P, Warms CA, Pelzer E, Rau H, Temkin N. Validity of the Patient Health Questionnaire-9 in assessing depression following traumatic brain injury. J Head Trauma Rehabil. 2005 Nov-Dec;20(6):501-11. doi: 10.1097/00001199-200511000-00003. PMID 16304487
- [Background] Ballesteros J, Santos B, Gonzalez-Fraile E, Munoz-Hermoso P, Dominguez-Panchon AI, Martin-Carrasco M. Unidimensional 12-item Zarit Caregiver Burden Interview for the assessment of dementia caregivers' burden obtained by item response theory. Value Health. 2012 Dec;15(8):1141-7. doi: 10.1016/j.jval.2012.07.005. Epub 2012 Oct 4. PMID 23244818
- [Derived] Juengst SB, Silva V, Goldin Y, Cicerone K, Lengenfelder J, Chiaravalloti N, Driver S, Mellick D, Dart G, Kew CL, Nabasny A, Bell KR. Care partner problem solving training (CP-PST) for care partners of adults with traumatic brain injury during inpatient rehabilitation: Study protocol for a multisite, randomized, single-blind clinical feasibility trial. Contemp Clin Trials. 2019 May;80:9-15. doi: 10.1016/j.cct.2019.03.004. Epub 2019 Mar 16. PMID 30885800
- Available data/document: Individual Participant Data Set: 602d — https://www.tbindsc.org/StaticFiles/SOP/602d%20-%20External%20Use%20TBIMS%20National%20Database%20Notification.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Solving Training + Education: Participants in this arm will receive the TBI-specific education intervention and the Problem Solving Training (PST) intervention.
  PST: This consists of six sessions that will follow a structured format based on the PST manual. The interventionist will first provide the TBI-specific education, introduce the participant to the PST steps, then help the care partner generate and select a problem to address first. Interventionist will facilitate the care partner's use of the ABCDEF steps of PST to develop a specific action plan to solve the problem. As problems are attempted or solved, care partner will learn how to perform the steps on his/her own, thus acquiring self-management problem solving skills that will be applicable to future problems. Final session will include a review and generalization of the PST steps and progress made.
  Education: Participants will receive TBI-specific education alone through a workbook. The modules consist of a brief introduction, key definitions, examples, resources, and a summary. Some chapters also include self-directed activities, such as worksheets or checklists. The investigators will provide a brief orientation to the workbook and include open-ended questions about the participants' need for clarification or questions of the education material. The last session will consist of an open discussion about expected problems that may arise post-discharge.
Period: Overall Study
Arm/Group | Problem Solving Training + Education | Education
Started | 43 | 51
Completed | 29 | 28
Not Completed | 14 | 23

BASELINE CHARACTERISTICS:
Population: n = 14 participants (n = 6 allocated to PST; n = 8 allocated to Education) who consented did not complete baseline assessment and no information is available for these participants. Therefore, of the 94 consented, baseline data are available for n=80 participants (n=37 PST, n=43 education only)
Groups:
- Problem Solving Training + Education: Participants in this arm will receive the TBI-specific education intervention and the Problem Solving Training (PST) intervention.
  Problem Solving Training (PST): The PST intervention consists of six sessions that will follow a structured format based on the PST manual. In these sessions, the interventionist will first provide the TBI-specific education, introduce the participant to the PST steps, then help the care partner generate and select a problem to address first. Interventionist will facilitate the care partner's use of the ABCDEF steps of PST to develop a specific action plan to solve the problem. As problems are attempted or solved, the care partner will learn how to perform the steps on his/her own, thus acquiring self-management problem solving skills that will be applicable to future problems. The final session will include a review and generalization of the PST steps and progress made.
  Education: Participants will receive TBI-specific education alone through a workbook. The modules consist of a brief introduction, key definitions, examples, resources, and a summary. Some chapters also include self-directed activities, such as worksheets or checklists. The investigators will provide a brief orientation to the workbook and include open-ended questions about the participants' need for clarification or questions of the education material. The last session will consist of an open discussion about expected problems that may arise post-discharge.
- Total: Total of all reporting groups
Arm/Group | Problem Solving Training + Education | Education | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.0) | 49.5 (15.7) | 49.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 65
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 20 | 36 | 56
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 4 | 1 | 5
Depression (Patient Health Questionnaire) [Mean (Standard Deviation); unit: units on a scale] — Population: The 1 participant in the Education arm did not complete the measure
  units on a scale
    number analyzed (Participants) | 37 | 42 | 79
    (all) | 8.6 (6.4) | 7.4 (5.3) | 7.96 (5.18)

OUTCOME MEASURES:

1. Primary Outcome: Changes From T2 to T3 in the Patient Health Questionnaire (PHQ9)
Description: The PHQ-9 assesses the frequency over the past two weeks of each of the nine symptoms of DSM-IV-TR that define a major depressive episode. Total scores range from 0-27, with established interpretative symptom cut-off scores of 0-4 (none), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and >20 (severe).(positive = improvement)
Time Frame: 1-month (T2), 6-month (T3) post-discharge between both arms
Population: The participants not analyzed here were lost to follow-up. These numbers do not match directly with the numbers in the participant flow since these are change scores. Therefore, participants had to have BOTH T2 and T3 data to be included in analysis.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Problem Solving Training + Education | Education
Number analyzed (Participants) | 11 | 17
change score on a scale | 2.9 (4.8) | 1.5 (3.2)

2. Primary Outcome: Changes T2 to T3 in the Zarit Burden Interview (ZBI) Group/Arm Differences at T2 in the ZBI
Description: The ZBI is a self-reported measure of perceived caregiver burden, including psychological health, well-being, social and family life, finances, and perceive control. There are multiple versions of the ZBI, but the investigators will use the 22-item version (each scored on a 5-pt Likert Scale), because it has been found to have good internal consistency reliability (α=.92) and established reference values for interpretation (mild: 2-20; mild to moderate: 21-40; moderate to severe:41-60; severe: 61-88). (positive = improvement)
Time Frame: 1 month (T2) and 6 month (T3) post-discharge between both arms
Population: The participants not analyzed here were lost to follow-up.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Problem Solving Training + Education | Education
Number analyzed (Participants) | 11 | 16
change score on a scale | 7.7 (10.4) | 2.6 (10.0)

3. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: The AUDIT is a 10-item screening tool for alcohol use behaviors designed by the World Health Organization to screen for alcohol abuse.The AUDIT assesses consumption, drinking behaviors, and alcohol-related problems. Scores range from 0-30, with a score of >8 indicating harmful alcohol use. Change scores were calculated from baseline to 6-month post-discharge.
Time Frame: Baseline and 6-month post-discharge
Population: Participants not included in analysis were lost to follow-up. These numbers do not directly align with numbers in the participant flow chart since analyses were planned for change scores, requiring data at BOTH time points.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Problem Solving Training + Education | Education
Number analyzed (Participants) | 17 | 22
change score on a scale | 0.59 (1.58) | 1.14 (2.38)

4. Secondary Outcome: Brief Coping Orientation to Problems Experienced
Description: The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The coping style of interest was Problem-Focused coping, with higher scores indicating more use of these kinds of coping strategies (higher scores are better; 8 items from the overall 28). Scores could range from 8 to 32. Differences scores were calculated for change from T2 to T3
Time Frame: 1-month (T2) and 6-month (T3) post-discharge
Population: Includes all participants with outcome data for this measure at both T2 and T3 (necessary to calculate change score). Participants not included were lost to follow-up at either or both time points.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Problem Solving Training + Education | Education
Number analyzed (Participants) | 11 | 11
change score on a scale | -1.00 (4.12) | 0.41 (5.21)

ADVERSE EVENTS:
Time Frame: From consent up to 6 months follow-up
Arm/Group | Problem Solving Training + Education | Education
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/51
Other Adverse Events (participants affected / at risk) | 0/43 | 0/51

LIMITATIONS AND CAVEATS:
In reviewing the original submitted protocol, the time frame of interest for a change in the primary and secondary outcome measures was 1 month to 6 months (all post-intervention), given the timing of the intervention delivery relative to onset of the care recipient's condition and the nature of the outcomes. This was a feasibility study to inform a future efficacy trial; decisions about timing, measures, and recruitment were the primary goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03739450/Prot_SAP_000.pdf